CLINICAL TRIAL: NCT07260864
Title: Investigating the Differential Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Left and Right Motor Cortex in Fibromyalgia: A Prospective Randomized Trial With Functional Magnetic Resonance Imaging (MRI(
Brief Title: Investigating the Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on the Brain in People With Fibromyalgia
Acronym: rTMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Paul Geha, Associate Professor of psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY0000010795; Schmitt program (Other Grant/Funding Number: URMC)
Record Dates: First submitted 2025-08-11; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia (FM)
Keywords: Transcranial Magnetic Stimulation; Chronic Pain; Nociplastic pain; Functional Magnetic Resonance Imaging; Motor Cortex
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Nociplastic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study will utilize single-blind as blinded outcome assessment, ensuring that investigators responsible for outcome evaluation and data analysis remain blinded to patients and whether treatment was delivered to the right or left motor cortex (M1). However, the clinician administering rTMS will not be blinded to the intervention arm (right vs left).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- right M1 rTMS (Active Comparator)
  Interventions: Other: rTMS
- Left M1 rTMS (Active Comparator)
  Interventions: Other: rTMS

INTERVENTIONS:
Other: rTMS — Using rTMS, which is a procedure that uses magnetic fields to stimulate nerve cells in the brain, to investigate its potential analgesic effects in fibromyalgia.

SUMMARY:
The first goal of this study is to see how brain activity changes in people with fibromyalgia after they get a treatment called rTMS (repetitive transcranial magnetic stimulation). Researchers are looking at how the parts of the brain that control movement (called motor cortices) respond to this treatment.

The second goal is to find out if the changes in brain activity are different between the right and left sides of the brain, depending on which side gets the treatment.

DETAILED DESCRIPTION:
The first aim of this study is to measure changes in fibromyalgia-related functional brain plasticity, as indicated by the functional "connectopy" of the right and left primary motor cortices in response to rTMS treatment. The second aim of this study is to explore whether changes in motor cortex connectopy differ between the right and left motor cortex (M1) following rTMS administered to each respective hemisphere.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 to 65, right-handed, with no racial/ethnic restrictions.
* A diagnosis of fibromyalgia by a qualified physician according to the American College of Rheumatology 2016 criteria
* Must have a history of fibromyalgia pain for a duration ≥ 3 months, as it is included in the diagnostic criteria.
* Must have pain intensity equal or greater than 4/10 on the numerical rating scale (NRS) at enrollment.
* Concurrent chronic overlapping pain conditions (except migraine with aura), depression, and anxiety will be allowed when mild to moderate (Less than 31 on Beck Depression Inventory or less than 36 on Beck Anxiety Inventory), except in cases with psychotic or manic features.
* Concomitant medication (except tricyclics, antipsychotic medications, bupropion, methadone, theophylline) and their doses for mood, pain and sleep disorders must be steady at least 4 weeks before enrolment and must be kept at a steady dosage during the trial.
* Must be able to read and speak English and be willing to read and understand instructions as well as questionnaires.
* Must be in generally stable health.
* Must sign an informed consent document after explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate.

Exclusion Criteria:

* Inability to provide informed consent.
* Age outside the studied range (i.e., < 18, > 65).
* Patients planning to change their medications during trial.
* Participants who are currently receiving other alternative therapies during trial (e.g., physiotherapy, acupuncture).
* History of receiving TMS, transcranial direct current stimulation (tDCS), or electroconvulsive therapy (ECT).
* Evidence of rheumatologic disorders, autoimmune diseases, taking immunosuppressive treatment, severe or unstable cardiac diseases.
* Fibromyalgia must be the primary complaint; hence patients cannot have another main source of pain (e.g., osteoarthritis). Patients will be asked to shade all the areas in which they experience pain on a body map. If they shade areas other than typical fibromyalgia pain, we will discuss any previous diagnosis, the intensity and chronicity of pain, and exclude them if chronic pain in any area outside the condition in to be studied is confirmed.
* Involvement in litigation regarding their pain or having a disability claim or receiving workman compensation or seeking either because of their pain.
* Any history of hemorrhagic or thrombotic stroke.
* History of schizophrenia, schizoaffective disorder, bipolar disorders, mania, hypomania, eating disorders, or any psychiatric illness with psychotic features (major depressive disorder, mild to moderate without psychosis, or anxiety disorders are not exclusion criteria).
* Current use of tricyclic antidepressants or any antipsychotic medications, given the risk of seizure incidence independent of TMS use in tricyclics is up to 0.4% or second-generation antipsychotics up to 1.2%.
* Significant other medical disease such as unstable diabetes mellitus, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, sleep apnea, or malignancy. Stable diabetes mellitus, stable hypertension (meaning that these conditions are followed up on by a physician and they are getting treatment for it with clinical stability), or hyperlipidemia are not exclusion criteria.
* History of traumatic brain injury
* History of epileptic disorders or family history of seizures in first degree relatives
* History of syncope
* History of tinnitus or hearing loss
* Current or history of substance misuse/dependence including alcohol at time of entry into the study.
* History of COVID-19 infection with persistent neurologic symptoms.
* Intra-axial implants (e.g., spinal cord stimulators or pumps) that are MRI incompatible.
* All exclusion criteria for MRI and TMS safety: any metallic implants, chips, or plates, cochlear implants, brain or skull abnormalities, aneurysm clips or coils, non-removable piercings, tattoos containing ferromagnetic ink, and claustrophobia.
* Surgery within the past 3 months or history of any brain surgery
* Pregnancy
* Participation into another research study
* In the judgment of the investigator, unable or unwilling to follow the protocol and instructions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Primary Motor Cortex (M1) Connectopy Profile | Baseline and post-treatment (after 10 sessions of rTMS over 2 weeks).
  Resting-state fMRI will be used to derive connectopy embeddings of the primary motor cortex (M1). Connectopy embeddings from the stimulated side will be extracted from significant baseline-defined clusters. A single value per participant is derived by averaging the embedding values within this cluster. Higher scores indicate increased similarity to healthy reference profiles (improved functional connectivity), while lower scores indicate deviation from healthy reference patterns (reduced functional connectivity).

SECONDARY OUTCOMES:
Mean Change in Pain Intensity (Numeric Rating Scale, NRS) | Baseline and post-treatment (following 10 rTMS sessions, within 7 days of completing rTMS sessions ).
  Self-reported average pain over 7 days using the Numeric Rating Scale (0 = "no pain at all" to 10 = "worst pain possible"). A single number is derived as the mean of daily ratings over 7 days. Lower scores indicate reduced pain intensity, while higher scores indicate worse pain intensity.
Mean Change in Pressure Pain Threshold (PPT) | Baseline and post-treatment (within 7 days of completing rTMS sessions )
  Pressure pain threshold (PPT) will be measured using a pressure algometer (Wagner Inc.). Pressure will be applied at a constant rate until participants indicate pain perception. The threshold (kg/cm²) will be recorded. A single value is derived by averaging three threshold readings from the target site. Higher thresholds indicate reduced pain sensitivity (improvement), while lower thresholds indicate increased pain sensitivity (worsening).
Mean Change in Fatigue (Patient-Reported Outcomes Measurement Information System-PROMIS Fatigue 13a Subscale) | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  Fatigue will be assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Fatigue 13a subscale, which ranges from 13 to 65. Higher scores indicate greater fatigue severity (worsening), whereas lower scores indicate less fatigue (improvement).
Mean Change in Sleep Disturbance (Patient-Reported Outcomes Measurement Information System - PROMIS Sleep Disturbance 8a Subscale) | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  Sleep disturbance will be assessed using the PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance 8a subscale, which ranges from 8 to 40. Higher scores indicate greater sleep disturbance (worsening), whereas lower scores indicate improved sleep.
Mean Change in the Short-Form McGill Pain Questionnaire | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) has 22 items assessing continuous, intermittent, neuropathic, and affective pain. Items are rated 0-10, with total scores ranging 0-220, where higher scores indicate greater pain severity.
Mean Change in Central Sensitization Index | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  Central Sensitization Index (CSI) is a 25-item self-reported measure that determines whether the symptoms of patients are associated with central sensitization. Item responses are on a 4-point scale and can be answered as follows: 0 = Never, 1 = Rarely, 2 = Sometimes, 3 = Often, and 4 = Always. The total score will be used to estimate the severity of the central sensitization symptoms.
Mean Change in Pain Catastrophizing Scale | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Pain Catastrophizing Scale (PCS) has 13 items measuring rumination, magnification, and helplessness related to pain. Items are rated 0-4, with total scores ranging 0-52; higher scores indicate greater catastrophizing.
Mean Change in the Pain Self-repot Survey for the Assessment of Fibromyalgia | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Patient Self-Report Survey for the Assessment of Fibromyalgia has 9 items measuring widespread pain and symptom severity. Scores range 0-31, with higher scores indicating greater fibromyalgia symptom burden.
Mean Change in Revised Fibromyalgia Impact Questionnaire | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Revised Fibromyalgia Impact Questionnaire (FIQR) is a 21-item, three-domain, self-reported measure of the impact of fibromyalgia on life. All questions include a 0-10 scale, and different domains have different calculations (function domain divided by 3, overall impact domain divided by 1, symptom domain divided by 2) before summing all scores. The total score will be used to estimate the changes in quality of life with interventions.
Mean Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Pittsburgh Sleep Quality Index (PSQI) measures sleep quality over the past month and consists of seven components assessing various aspects of sleep quality and sleep-related daytime functioning. The index will be used to estimate the overall sleep quality of participants, with total scores ranging from 0 to 21, where higher scores indicate worse sleep quality.
Mean Change in Chronic Overlapping Pain Conditions Screener | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  Chronic Overlapping Pain Conditions Screener (COPCS) is a self-report tool that uses a body map and trigger questions to screen for 10 chronic overlapping pain conditions and outputs the number of conditions present (0-10).
Mean Change in Hospital Anxiety and Depression Scale | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Hospital Anxiety and Depression Scale (HADS) has 14 items, 7 each for anxiety and depression. Each item is rated 0-3, with subscale scores ranging 0-21; higher scores indicate greater symptom severity.
Mean Change in Beck Depression Inventory | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Beck Depression Inventory (BDI) has 21 items assessing depressive symptoms. Each item is rated 0-3, with total scores ranging 0-63; higher scores indicate greater depression severity.
Mean Change in Beck Anxiety Inventory | Baseline and post-treatment (within 7 days of completing rTMS sessions).
  The Beck Anxiety Inventory (BAI) has 21 items assessing anxiety symptoms. Each item is rated 0-3, with total scores ranging 0-63; higher scores indicate greater anxiety severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No